CLINICAL TRIAL: NCT01885156
Title: A Phase 3 Double-Blind, Randomized, Placebo-Controlled, Multicenter, Parallel Group Evaluation of the Efficacy and Safety of Naftin 1% Cream in Adolescent Subjects With Tinea Cruris
Brief Title: Evaluation of Efficacy and Safety of Naftin 1% Cream in Adolescent Subjects With Tinea Cruris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MUS 90200_3028_1
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-03

CONDITIONS: Tinea Cruris; Jock Itch
MeSH Terms: conditions — Tinea Cruris | interventions — naftifine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Cream (Placebo Comparator): Topically applied once daily
  Interventions: Drug: Placebo Cream
- Naftin 1% Cream (Experimental): Topically applied once daily
  Interventions: Drug: Naftin 1% Cream

INTERVENTIONS:
Drug: Naftin 1% Cream — Topically applied once a day
  Arms: Naftin 1% Cream
Drug: Placebo Cream — Topically applied once a day
  Arms: Placebo Cream

SUMMARY:
To see how well Naftin 1% cream works when applied once daily to the affected area. The results will be compared to those using a placebo cream, which is a cream with no active ingredient. Safety will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Review and sign statement of Informed Consent and HIPAA authorization.
* Males or non-pregnant females ≥ 12 years of age to 17 years, 11 months, of any race or sex. Females of child-bearing potential must have a negative urine pregnancy test.
* The parent/legal guardian must complete the informed consent process AND the subject must complete the assent process and sign the appropriate form (if age appropriate).
* Presence of tinea cruris characterized by clinical evidence of a tinea infection (at least moderate erythema, moderate scaling, and mild pruritus) based on signs and symptoms.
* KOH positive baseline skin scrapings obtained from the site most severely affected or a representative site of the overall severity.
* Subjects must be in good health and free from any clinically significant disease that might interfere with the study evaluations.
* Subject must be able to understand the requirements of the study and willing to comply with the study requirements.

Exclusion Criteria:

* A life threatening condition (ex. autoimmune deficiency syndrome, cancer, unstable angina, or myocardial infarction) within the last 6 months.
* Subjects with abnormal findings - physical or laboratory - that are considered by the investigator to be clinically important and indicative of conditions that might complicate interpretation of study results.- Severe dermatophytoses, mucocutaneous candidiasis, or bacterial skin infection.
* Subjects with a known hypersensitivity to study medications or their components.
* Subjects who have a recent history or who are currently known to abuse alcohol or drugs.
* Uncontrolled diabetes mellitus.
* Hemodialysis or chronic ambulatory peritoneal dialysis therapy.
* Current diagnosis of immunocompromising conditions.
* Atopic or contact dermatitis.
* Severe dermatophytoses, mucocutaneous candidiasis, or bacterial skin infection.
* Female subject who is pregnant or lactating, who is not using or does not agree to use an acceptable form of contraception during the study, or who intends to become pregnant during the study (females who are surgically sterilized for at least 2 years are not considered to be of childbearing potential).
* Subjects using the following medications:

  * Topical anti-fungal therapy, powders or topical corticosteroids applied within 14 days prior to randomization. Terbinafine, butenafine, and naftifine (topical) within 30 days prior to randomization.
  * Oral anti-fungal therapies within 3 months of randomization (8 months for oral terbinafine).
  * Systemic antibiotic or corticosteroid treatment within 30 days of randomization.
  * Any other significant treatments, except hormonal contraception and multivitamin, at the discretion of the investigator that would interfere with study treatment.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Safety of Naftin® 1% Cream, applied once daily for 4 weeks, compared to vehicle for treatment of subjects with KOH positive symptomatic tinea cruris in adolescent subjects (aged 12 years to 17 years, 11 months). | Week 6
  - Summarization of AEs (local and systemic)

SECONDARY OUTCOMES:
Efficacy of Naftin® 1% Cream, applied once daily for 4 weeks, compared to vehicle for treatment of subjects with KOH and culture positive symptomatic tinea cruris in adolescent subjects (aged 12 years to 17 years, 11 months). | Week 6
  Complete Cure based on:
  -Negative mycology results; absence (Grade 0) of erythema, scaling, and pruritis
  Other efficacy variables assessed at Week 2, Week 4, and Week 6:
  * Effective treatment
  * Mycological cure
  * Clinical Success
  * Clinical Cure
  * Investigator Global Assessment
  * Subject Satisfaction Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Plaum, MD, Study Director — Merz North America, Inc.
Locations (5):
- Belize (2):
  - Merz Investigational Site # 501001, Belize City
  - Merz Investigational Site # 501002, Belize City
- Dominican Republic (2):
  - Merz Investigative Site # 180002, San Cristóbal
  - Merz Investigative Site # 180001, Santo Domingo
- Merz Investigative Site # 504001, San Pedro Sula, Honduras